CLINICAL TRIAL: NCT01571739
Title: Risk Stratification in Latent Tuberculosis: PET/CT Findings in TB Contacts
Brief Title: Determining Risk in Latent Tuberculosis
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912036; 12-I-N036
Record Dates: First submitted 2012-04-04; First posted 2012-04-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2014-05-20

CONDITIONS: Latent Tuberculosis
Keywords: Biomarker; Latent Tuberculosis; IGRA; Isoniazid; TB Lymphadenopathy; Tuberculosis; TB
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Tuberculosis (TB) is a leading cause of death worldwide. Those who are exposed to the TB bacteria but have not become sick are said to have latent TB. Many people with latent TB will not get sick from it, but some people will develop active TB and become sick. Much is known about how to treat and diagnose active TB, but little is known about the best way to treat latent TB. Researchers also want to know more about the risk that latent TB will develop into active TB, and whether it is possible to test for this risk.

Objectives:

- To test possible methods of determining a person s risk for developing active TB.

Eligibility:

- Individuals between 20 and 60 years of age who (1) have active TB, (2) were exposed to someone with active TB in the past 9 months, or (3) have not been exposed to TB.

Design:

* Participants will be separated into groups based on their exposure to TB.
* Healthy participants who were not exposed to TB will answer questions about their medical history. They will also provide blood and urine samples.
* Participants who have active TB will have a physical exam and medical history. They will provide blood, urine, and sputum samples, and will have a chest x-ray. They will be treated with the standard of care for active TB. Some participants with active TB may have additional tests as part of this study.
* Participants who were exposed to TB and have latent TB will have a physical exam and medical history. They will provide blood, urine, and sputum samples, and will have a chest x-ray. They will be asked to return for five more clinic visits over the next 12 months to repeat these tests. They may also have additional chest imaging studies depending on the study needs.
* Some of the exposed participants may have been exposed to drug-resistant TB. These participants will receive the drug isoniazid to take on a regular schedule to help prevent the latent TB from becoming active TB.

DETAILED DESCRIPTION:
The efficacy of treating tuberculin skin test (TST) positive, or interferon gamma release assay (IGRA) positive, contacts of tuberculosis (TB) cases to prevent progression to disease is well established. However the length of treatment, and the toxicity associated with the currently used regimens, means that the risk may outweigh the benefit and treatment completion rates are poor. In addition, no proven regimens are available for contacts of multidrug resistant tuberculosis (MDR-TB) cases. Because as few as 2% of contacts develop active TB over 1 year and no surrogate markers are available, drug trials to assess novel treatments typically require thousands of subjects followed up for many years. (18F)-fluoro-2-deoxy-D-glucose positron emission tomography/computer tomography (FDG-PET/CT) may prove a useful surrogate for more targeted chemoprophylaxis as well as a means to rapidly evaluate novel prophylactic regimes in future studies.

Up to 40% of immune-sensitized TB contacts with normal chest radiographs (CXR) have abnormalities on conventional chest CT. FDG-PET/CT not only will allow characterization of the metabolic activity of these lesions but is also likely to reveal significantly increased metabolic activity within regional lymph nodes that may otherwise be anatomically normal. Based on previous studies, we predict that up to 65% of contacts will have combined chest PET/CT abnormalities and that up to 50% of contacts who are treated, will have increased FDG uptake that will resolve with treatment. By contrast, PET screening studies demonstrate abnormal pulmonary FDG uptake occurs in 0.9% of healthy individuals.

The development of biomarkers more predictive of disease progression is also highly desirable, but for similar reasons evaluating them is challenging. This novel approach of using FDG-PET/CT to benchmark the dynamic immunological, transcriptional, or metabolic changes that occur early in tuberculosis infection, we hope will accelerate biomarker discovery. In this study we propose to evaluate these predictions in order to lay the foundation for future studies.

ELIGIBILITY:
* INDEX CASES:

INCLUSION CRITERIA:

1. Either confirmed sputum smear positive and culture positive for M. tb within the last 12 months OR sputum smear positive and genotypically confirmed M.tb with culture awaited
2. Age greater than or equal to 20 years old

20 Smear Positive Pulmonary TB Biomarker Index Case Controls:

INCLUSION CRITERIA:

1. Genotypically confirmed sputum smear positive pulmonary tuberculosis
2. Culture awaited or confirmed Mtb
3. Not commenced anti-tuberculous therapy
4. Age greater than or equal to 20 years old

EXCLUSION CRITERIA:

1. Age >60 years old
2. Known diagnosis of chronic inflammatory condition (e.g. Sarcoid, RA, connective tissue disorder) or on immunosuppressive medication

WITHDRAWAL CRITERIA:

1) Culture negative for M.tb

QF-GIT Positive Contacts:

INCLUSION CRITERIA:

1. Contacts of index case
2. QF-GIT positive
3. Age greater than or equal to 20 years old
4. Normal CXR

EXCLUSION CRITERIA:

1. Exposure to an index case who commenced treatment for a current episode of TB (one that was not successfully treated, per WHO definition) more than 15 months ago
2. Previously diagnosed or treated TB
3. Symptoms or signs of active TB
4. Symptoms or signs of acute illness
5. CXR suggestive of active tuberculosis or parenchymal abnormalities known or suspected to be caused by alternative pathology
6. HIV positive or other significant immunocompromise
7. Age >60
8. Smoker >30 pack years
9. Previously diagnosed malignancy
10. Previously diagnosed chronic lung infection (e.g., non tuberculosis mycobacteria [NTM], Fungal, Paragonimus)
11. Known diagnosis of chronic inflammatory condition associated with pulmonary pathology (e.g., Sarcoidosis, RA, Wegener s granulomatosis, bronchiectasis)
12. Inhaled or systemic steroid use within previous 2 weeks (subject may return for enrollment 2 weeks after last dose) and need for ongoing steroid therapy
13. Breast feeding, pregnant, or planning pregnancy
14. Anticipated poor compliance

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01-02; Study Completion 2014-05-20

PRIMARY OUTCOMES:
To estimate the rate of PET plus CXR at baseline among all study participants.

SECONDARY OUTCOMES:
To estimate the rate of PET+/CT- at baseline among all study participants.
To estimate the rate of regression of PET plus scans (to normal) at 3 and 12 months among the untreated subjects (n=30).

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Banura C, Mirembe FM, Katahoire AR, Namujju PB, Mbonye AK, Wabwire FM. Epidemiology of HPV genotypes in Uganda and the role of the current preventive vaccines: A systematic review. Infect Agent Cancer. 2011 Jul 12;6(1):11. doi: 10.1186/1750-9378-6-11. PMID 21749691
- [Background] Block SL, Nolan T, Sattler C, Barr E, Giacoletti KE, Marchant CD, Castellsague X, Rusche SA, Lukac S, Bryan JT, Cavanaugh PF Jr, Reisinger KS; Protocol 016 Study Group. Comparison of the immunogenicity and reactogenicity of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in male and female adolescents and young adult women. Pediatrics. 2006 Nov;118(5):2135-45. doi: 10.1542/peds.2006-0461. PMID 17079588
- [Background] Centers for Disease Control and Prevention (CDC). National, state, and local area vaccination coverage among adolescents aged 13-17 years --- United States, 2009. MMWR Morb Mortal Wkly Rep. 2010 Aug 20;59(32):1018-23. PMID 20724968